CLINICAL TRIAL: NCT05847673
Title: Avatar-Led Digital Therapeutic to Aid Smoking Cessation Among Sexual and Gender Minority Young Adults
Brief Title: Avatar-Led Digital Therapeutic for Aiding Smoking Cessation in Sexual and Gender Minority Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: The Leonard and Norma Klorfine Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RG1123270; NCI-2023-03050 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1123270 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Smoking Devices; Health Promotion; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (EQQUAL A) (Experimental): Participants receive self-guided online EQQUAL A program on study. Participants also receive motivational messages and smoking cessation information via text messages.
  Interventions: Behavioral: Online Smoking Cessation Intervention; Other: Questionnaire Administration; Other: Health Promotion and Education
- Arm II (EQQUAL B) (Active Comparator): Participants receive self-guided online EQQUAL B program on study. Participants also receive motivational messages and smoking cessation information via text messages.
  Interventions: Behavioral: Online Smoking Cessation Intervention; Other: Questionnaire Administration; Other: Health Promotion and Education

INTERVENTIONS:
Behavioral: Online Smoking Cessation Intervention — Receive EQQUAL A intervention
  Other Names: Smoking and Tobacco Use Cessation Intervention
  Arms: Arm I (EQQUAL A)
Behavioral: Online Smoking Cessation Intervention — Receive EQQUAL B intervention
  Other Names: Smoking and Tobacco Use Cessation Intervention
  Arms: Arm II (EQQUAL B)
Other: Questionnaire Administration — Ancillary studies
Other: Health Promotion and Education — Receive motivational messages and smoking cessation information via SMS text messages

SUMMARY:
This trial assesses the acceptability and preliminary efficacy of Empowered, Queer, Quitting, and Living (EQQUAL) smoking-cessation intervention for sexual and gender minority young adult smokers. The prevalence of tobacco use among sexual and gender minority (SGM) young adults is more than twice as high as non-SGM young adults, suggesting that existing SGM-related disparities in tobacco use will persist well into the foreseeable future unless sustained efforts are undertaken to address them. EQQUAL is an online smoking cessation intervention designed specifically for SGM young adult smokers, and may help them quit smoking.

DETAILED DESCRIPTION:
OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive self-guided, online quit smoking program, called EQQUAL Program A.

ARM II: Participants receive self-guided online quit smoking program, EQQUAL Program B.

ELIGIBILITY:
Inclusion Criteria:

* DEMOGRAPHIC CRITERIA:
* Participants must self-identify being between 18 and 30 years of age
* Participants must self-identify as a sexual and/or gender minority (i.e., a sexual orientation other than straight and/or gender that doesn't match sex assigned at birth)
* Participants must currently reside in the United States, with a United States (US) mailing address, and anticipate remaining in the US for the duration of the study (3 months)
* SMOKING CRITERIA:
* Participants must self-report smoking at least 1 cigarette per day in the 30 days prior to screening
* TREATMENT ACCESSIBILITY:
* Participants must self-report having at least weekly Internet access for the next three months
* Participants must self-report being willing and able to stream audio and video online for this study
* Participants must self-report current use of a personal email account
* Participants must self-report current use of text messaging
* OTHER CRITERIA:
* Participants must self-report that they are interested in participating in the study for themselves (versus [vs] someone else)
* Participants must self-report that they have not participated in one of our prior smoking cessation studies
* Participants must self-report that they are comfortable reading, writing, and speaking English
* Participants must self-report that they understand and agree to the conditions of compensation
* Participants must self-report that they are not currently incarcerated
* Participants must be willing to use the assigned intervention program, complete the study assessments, and consent to participate in this study
* Participants must be willing to upload a photo of themselves (face visible)

Exclusion Criteria:

* Participants must not be currently using other tobacco cessation treatments at the time of screening, including pharmacotherapy or behavioral support (but initiating these treatments during the study is allowed)
* Participants must not be a member of the same household as another research participant
* Having a Google voice number as their sole phone number

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Overall satisfaction | At 3-month follow-up
  Will be assessed with a 5-point Likert-type item on the 3-month survey. Responses will be recorded into a binary variable representing responses of "mostly satisfied" or "very satisfied" versus all other responses (i.e., "not at all," "a little," and "somewhat"). Will test for statistical differences between arms using a logistic regression, with adjustment for the stratification variables, as well as adjustment for any baseline variables that had a statistically significant difference by study arm and were associated with the outcome (i.e., potential confounders).
Average change in Contemplation Ladder scores | Baseline through 3-month follow-up
  Contemplation Ladder scores will be used to assess readiness to quit using cigarettes. Will test for statistical differences between arms using linear regression, with adjustment for the stratification variables, as well as adjustment for any baseline variables that had a statistically significant difference by study arm and were associated with the outcome (i.e., potential confounders).
Reduction in cigarettes smoked per day | Baseline through 3-month follow-up
  Change in cigarette smoked per day will be assessed as the difference between average number of cigarettes smoked per day over the past 7 days at baseline and at 3-month follow-up. Will test for statistical differences between arms using a negative binomial regression with adjustment for the stratification variables, as well as adjustment for any baseline variables that had a statistically significant difference by study arm and were associated with the outcome (i.e., potential confounders).
7-day point prevalence abstinence (PPA) from all nicotine and tobacco use | At 3-month follow-up
  Self-report of no nicotine and tobacco use over the past 7 days, biochemically confirmed via saliva cotinine. Will test for statistical differences between arms using a logistic regression, with adjustment for the stratification variables, as well as adjustment for any baseline variables that had a statistically significant difference by study arm and were associated with the outcome (i.e., potential confounders).
Usability of the Empowered, Queer, Quitting, and Living (EQQUAL) program | At 3-month follow-up
  Measured by the System Usability Scale. Will be presented descriptively as an average usability score.
Acceptability of the EQQUAL avatar | At 3-month follow-up
  Will be assessed using the Agent Persona Instrument, an adapted version of the Robotics Social Attribute Scale, and 4 open-ended, study specific questions. Will be presented descriptively as frequencies and percentages.
Number of EQQUAL sessions completed | Up to 3 months
  Will be presented descriptively as frequencies and percentages.

SECONDARY OUTCOMES:
Changes in the acceptance of smoking triggers | Baseline through 3-month follow-up
  Assessed by the emotional and physical subscales of the Avoidance and Inflexibility Scale (AIS). Will calculate the change score as 3-month follow-up minus baseline score and use a linear regression model with adjustment for the baseline value of the measure of interest and for the stratification variables, as well as adjustment for any baseline variables that had a statistically significant difference by study arm and were associated with the outcome.
Changes in psychological flexibility | Baseline through 3-month follow-up
  Assessed by the short version of the Multidimensional Psychological Flexibility Inventory (MPFI). Will calculate the change score as 3-month follow-up minus baseline score and use a linear regression model with adjustment for the baseline value of the measure of interest and for the stratification variables, as well as adjustment for any baseline variables that had a statistically significant difference by study arm and were associated with the outcome.
Changes in valued living | Baseline through 3-month follow-up
  Assessed by the Valuing Questionnaire. Will calculate the change score as 3-month follow-up minus baseline score and use a linear regression model with adjustment for the baseline value of the measure of interest and for the stratification variables, as well as adjustment for any baseline variables that had a statistically significant difference by study arm and were associated with the outcome.
Differences in 3-month smoking outcomes between those with high versus low baseline readiness to quit | Baseline through 3-month follow-up
  Will be presented descriptively as frequencies and percentages.
Differences in 3-month smoking outcomes between those who identify as gender minority versus those who don't | Baseline through 3-month follow-up
  Will be presented descriptively as frequencies and percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Jaimee Heffner, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT05847673/ICF_000.pdf